CLINICAL TRIAL: NCT02330380
Title: Comparative Effectiveness of Psoriasis Treatments on Systemic Inflammation
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Psoriasis Foundation (Other)
Responsible Party: Principal Investigator, Neil Korman, Principal Investigator, University Hospitals Cleveland Medical Center
Other Study IDs: 04-13-21
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Psoriasis; Inflammation
Keywords: psoriasis, comparative effects, inflammation
MeSH Terms: conditions — Psoriasis; Inflammation | interventions — Methotrexate; Ustekinumab; Etanercept; Adalimumab; Acitretin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies and blood samples will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Methotrexate: Methotrexate will be dosed weekly. Methotrexate is given as a single, weekly dose and is will be started at 15mg after a first week test dose of 2.5 mg to minimize side effects and achieve efficacy. Weekly dosages will be 15mg.
  Interventions: Drug: Methotrexate
- Ustekinumab: Ustekinumab is given as a subcutaneous injection of 45mg if the patient is <100Kg or 90mg if the patient is >100Kg at weeks 0, 4, 16, and every 12 weeks thereafter.
  Interventions: Drug: Ustekinumab
- Etanercept: Etanercept will be given in the first 3 months of treatment as 50 mg twice a week (3 or 4 days apart). After 3 months, a reduced dose of 50 mg will be given once per week.
  Interventions: Drug: Etanercept
- Adalimumab: Adalimumab will be given in a dose of 40 mg subcutaneously every other week.
  Interventions: Drug: Adalimumab
- Acitretin: Acetretin will be prescribed as daily with 25mg if the patient is <80Kg or 35mg if the patient is >80Kg.
  Interventions: Drug: Acitretin
- UVB Excimer Laser: Dose determination will be determined by a physician per standard-of-care by performing a Sunburn Test/Minimal Erythemal Dose Test, or by visually evaluating the patient's skin type and thickness of psoriasis plaque. Initial laser dose will be 1-4X the MED depending on the thickness of the plaque. Escalation will be 25-50% increase in dose per treatment if there is no residual erythema, 25% increase per treatment if there is mild residual erythema, and 0% increase per treatment if there is moderate residual erythema. Investigators also have the option to skip a treatment, if there is above moderate erythema, or significant patient discomfort. Patients will receive treatment twice a week.
  Interventions: Other: UVB Excimer Laser
- Narrowband UVB: Narrowband UVB (311nm) will be used to treat patients 3X per week with 311nm of UVB light. Uninvolved areas of skin will be covered where possible to minimize excess sun exposure. Patients will be tested for their minimal erythemal dose (MED), after which, based upon Fitzpatrick Scale skin type, a patient will typically beginning with 1-2 minutes based on skin type and gradually increased by 10-15% per treatment dose as tolerated.
  Interventions: Other: Narrowband UVB

INTERVENTIONS:
Drug: Methotrexate — Subjects will receive Methotrexate as detailed in the "Group" description.
  Groups: Methotrexate
Drug: Ustekinumab — Subjects will receive Ustekinumab as detailed in the "Group" description.
  Groups: Ustekinumab
Drug: Etanercept — Subjects will receive Etanercept as detailed in the "Group" description.
  Groups: Etanercept
Drug: Adalimumab — Subjects will receive Adalimumab as detailed in the "Group" description.
  Groups: Adalimumab
Drug: Acitretin — Subjects will receive Acitretin as detailed in the "Group" description.
  Groups: Acitretin
Other: UVB Excimer Laser — Subjects will receive UVB Excimer Laser therapy as detailed in the "Group" description.
  Groups: UVB Excimer Laser
Other: Narrowband UVB — Subjects will receive Narrowband UVB as detailed in the "Group" description.
  Groups: Narrowband UVB

SUMMARY:
This is a prospective longitudinal observational pilot study of psoriasis patients on continuous standard-of-care systemic therapeutics to determine the level of change in established (plasma/serum) and investigative (cellular) biomarkers that are associated with increased risk of CVD events.

The final endpoint of the proposed study will be a ranking of the examined biomarkers based upon an integrated assessment of biomarker behavior over time.

Secondary outcomes will assess changes in coronary artery calcification scoring, PET-MRI, skin biopsies, and clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 18-65 years old
* Diagnosis of moderate-to-severe plaque psoriasis
* Plaque affects ≥ 10% of subject's body surface area (BSA)
* Subjects prescribed one of the following standard-of-care treatments for their psoriasis: Ustekinumab, Methotrexate, Etanercept, Adalimumab, Narrow Band UVB (311nm), Excimer Laser Treatment (308nm), or Acitretin
* Subjects willing to complete a Washout Period prior to Visit 1 (only for subjects currently on a psoriasis treatment):

  * Discontinue systemic therapies for at least 4 weeks
  * Discontinue topical therapies for at least 2 weeks
  * Discontinue phototherapies for at least 2 weeks

Exclusion Criteria:

* Subjects who are currently on a psoriasis treatment and unwilling to go through the washout-period
* Subjects with a critical illness or who are immunocompromised
* Weight is 400lbs or greater
* Subjects who are currently pregnant or breastfeeding
* Subjects who have metal implants
* Subjects who have a pacemaker, stent, or artificial heart valve
* History of clinically significant hematological, renal or liver disease
* Patients with known co-morbidities that raise biomarkers such as:

  * History of myocardial infarction (MI)
  * History of cerebrovascular accident (CVA)
  * Significant atherosclerosis (defined as the presence of any carotid plaque; or carotid intimal media thickness (cIMT) >75th percentile for age; or the presence of coronary artery calcium score>100)
  * Poorly controlled diabetes (elevated HbA1c > 8.5)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psoriasis patients
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Biomarker assessment | 52 weeks
  The biomarkers examined throughout the study will be assessed. And, an integrated assessment of biomarker behavior over time will be performed. Biomarkers examined will include High sensitivity C-reactive protein (hsCRP), Myeloperoxidase (MPO), resistin, adiponectin and leptin.

SECONDARY OUTCOMES:
Changes in coronary artery calcification scoring | 52 weeks
  Coronary Artery Calcification Scoring (CACS) will be performed at the first and final visits for the study.
Changes in PET-MRI | 52 weeks
  Patients who enroll in this study will receive two PET/MRI scans. The first one will be done prior to beginning their psoriasis therapy during Visit 1 and the second PET/MRI will be done during the Final Visit.
Clinical improvement | 52 weeks
  Psoriasis Area Severity Index (PASI) and Static Physician Global Assessment (sPGA) will be performed throughout the study to monitor clinical improvement.
Changes in skin biopsies | 52 weeks
  In some patients, two 4-6mm punch biopsies will be obtained after the washout period has been observed, one from a psoriasis lesion and one from an adjacent, uninvolved area. Two 4-6mm punch biopsies will also be obtained during the final visit, one from a psoriasis lesion and one from an adjacent, uninvolved area.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Korman, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Alora-Palli MB, Brouda I, Green B, Kimball AB. A cost-effectiveness comparison of liquor carbonis distillate solution and calcipotriol cream in the treatment of moderate chronic plaque psoriasis. Arch Dermatol. 2010 Aug;146(8):919-22. doi: 10.1001/archdermatol.2010.167. No abstract available. PMID 20713833
- [Background] Ho SG, Yeung CK, Chan HH. Methotrexate versus traditional Chinese medicine in psoriasis: a randomized, placebo-controlled trial to determine efficacy, safety and quality of life. Clin Exp Dermatol. 2010 Oct;35(7):717-22. doi: 10.1111/j.1365-2230.2009.03693.x. PMID 19925489
- [Background] Flytstrom I, Stenberg B, Svensson A, Bergbrant IM. Methotrexate vs. ciclosporin in psoriasis: effectiveness, quality of life and safety. A randomized controlled trial. Br J Dermatol. 2008 Jan;158(1):116-21. doi: 10.1111/j.1365-2133.2007.08284.x. Epub 2007 Nov 6. PMID 17986302
- [Background] Heydendael VM, Spuls PI, Opmeer BC, de Borgie CA, Reitsma JB, Goldschmidt WF, Bossuyt PM, Bos JD, de Rie MA. Methotrexate versus cyclosporine in moderate-to-severe chronic plaque psoriasis. N Engl J Med. 2003 Aug 14;349(7):658-65. doi: 10.1056/NEJMoa021359. PMID 12917302
- [Background] Reich K, Sinclair R, Roberts G, Griffiths CE, Tabberer M, Barker J. Comparative effects of biological therapies on the severity of skin symptoms and health-related quality of life in patients with plaque-type psoriasis: a meta-analysis. Curr Med Res Opin. 2008 May;24(5):1237-54. doi: 10.1185/030079908x291985. Epub 2008 Mar 19. PMID 18355421
- [Background] Atteno M, Peluso R, Costa L, Padula S, Iervolino S, Caso F, Sanduzzi A, Lubrano E, Del Puente A, Scarpa R. Comparison of effectiveness and safety of infliximab, etanercept, and adalimumab in psoriatic arthritis patients who experienced an inadequate response to previous disease-modifying antirheumatic drugs. Clin Rheumatol. 2010 Apr;29(4):399-403. doi: 10.1007/s10067-009-1340-7. PMID 20066450
- [Background] Saurat JH, Stingl G, Dubertret L, Papp K, Langley RG, Ortonne JP, Unnebrink K, Kaul M, Camez A; CHAMPION Study Investigators. Efficacy and safety results from the randomized controlled comparative study of adalimumab vs. methotrexate vs. placebo in patients with psoriasis (CHAMPION). Br J Dermatol. 2008 Mar;158(3):558-66. doi: 10.1111/j.1365-2133.2007.08315.x. Epub 2007 Nov 28. PMID 18047523
- [Background] Mehta NN, Yu Y, Saboury B, Foroughi N, Krishnamoorthy P, Raper A, Baer A, Antigua J, Van Voorhees AS, Torigian DA, Alavi A, Gelfand JM. Systemic and vascular inflammation in patients with moderate to severe psoriasis as measured by [18F]-fluorodeoxyglucose positron emission tomography-computed tomography (FDG-PET/CT): a pilot study. Arch Dermatol. 2011 Sep;147(9):1031-9. doi: 10.1001/archdermatol.2011.119. Epub 2011 May 16. PMID 21576552
- [Background] Gelfand JM, Wan J, Callis Duffin K, Krueger GG, Kalb RE, Weisman JD, Sperber BR, Stierstorfer MB, Brod BA, Schleicher SM, Bebo BF Jr, Troxel AB, Shin DB, Steinemann JM, Goldfarb J, Yeung H, Van Voorhees AS. Comparative effectiveness of commonly used systemic treatments or phototherapy for moderate to severe plaque psoriasis in the clinical practice setting. Arch Dermatol. 2012 Apr;148(4):487-94. doi: 10.1001/archdermatol.2012.370. PMID 22508874